CLINICAL TRIAL: NCT05774418
Title: Evaluation of the Effectiveness and Safety of the BNT162b2 COVID-19 Vaccine in the Vaccination Campaign Among the Health Workers of Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Brief Title: Evaluation of the Impact of the Anti COVID-19 Vaccination Campaign Addressed to the Employees of an Italian Hospital.
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3973
Record Dates: First submitted 2023-03-13; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- vaccinated: Healthcare workers (aged ≥18 years) working at hospital sites who could provide written informed consent and who will complete the immunization program with the administration of the second dose after approximately 21 days from the first dose at the FPG
  Interventions: Biological: BNT162b2 COVID-19 Vaccine
- unvaccinated: unvaccinated health workers

INTERVENTIONS:
Biological: BNT162b2 COVID-19 Vaccine — BNT162b2 is a vaccine for preventing coronavirus disease 2019 (COVID-19) in people from the age of 18 years. BNT162b2 contains tozinameran, a messenger RNA (mRNA) molecule with instructions for producing a protein from the original strain of SARS-CoV-2, the virus that causes COVID-19. BNT162b2 is given as two injections, usually into the muscle of the upper arm, 3 weeks apart.
  Groups: vaccinated

SUMMARY:
Health workers, especially those in patient-facing roles, had a significantly increased risk of COVID-19 infection, having serious outcomes, and risking spreading the virus to patients and staff. Vaccination campaign planning suggests allocating initial supplies of BNT162b2 vaccine to health workers given the importance of early protection to safeguard the continuity of care to patients. The aim of the study is to assess the effectiveness and safety of BNT162b2 vaccine among the health workers of Fondazione Policlinico Universitario Agostino Gemelli IRCCS (FPG). The retrospective cohort study will be conducted among health staff working at the FPG. Vaccination data will collect from hospital records. The primary end points will be vaccine effectiveness and safety.

DETAILED DESCRIPTION:
On 11 March 2020, the rapidly spreading novel coronavirus outbreak was declared a pandemic by the World Health Organization (WHO). From that moment on, SARS-CoV-2 has affected hundreds of millions of people globally. As of 24 September 2021, as reported by the WHO, there have been 230,418,451 confirmed cases of COVID-19, including 4,724,876 deaths, worldwide. To date, the scientists reported that COVID-19 pandemic had a substantial burden of disease worldwide.

As an action to curb the burden of COVID-19, Italy authorized the marketing of Pfizer-BioNTech (BNT162b2) vaccine and licensed it for use after it showed high effectiveness and safety against symptomatic infection in a large multinational clinical trial. BNT162b2 is a lipid nanoparticle-formulated, nucleoside-modified RNA vaccine encoding a prefusion-stabilized, membrane-anchored SARS-CoV-2 full-length spike protein. In December 2020, Italy, jointly with other European countries, started the COVID-19 mass vaccination campaign, initially addressed to health workers, staff, and patients of homes for elderly people. Health workers, especially those in patient-facing roles, had a significantly increased risk of COVID-19 infection, having serious outcomes, and risking spreading the virus to patients and staff . Therefore, health workers have been prioritized to receive COVID-19 vaccines in many countries. By the end of March 2021, in the majority of the Italian hospitals, most health workers received both doses of the BNT162b2 COVID-19 vaccine, while few received both doses of mRNA-1273 (i.e., Moderna). In Italy, as of 25 September 2021, a total of 83,662,989 vaccine doses were administered, vaccinating 77.4% of the population aged over 12. As highlighted by the WHO , COVID-19 vaccines have been proven as safe, effective, and life-saving against this severe disease in several large vaccine trials. Several studies have been conducted to assess the effectiveness of vaccination campaigns in the health care workers in real-world settings. We add to this evidence by providing an assessment of the effectiveness and safety of (BNT162b2) vaccine among the health workers of Fondazione Policlinico Universitario Agostino Gemelli IRCCS (FPG), a large teaching hospital in Rome (Italy).

A retrospective cohort study among health staff working at the FPG will be conducted to evaluate the effectiveness and safety of BNT162b2 vaccine during the first phase of the vaccination campaign against SARS-CoV-2.

Healthcare workers (aged ≥18 years) working at hospital sites who could provide written informed consent and who will complete the immunization program with the administration of the second dose after approximately 21 days from the first dose at the FPG will be included.

Participants will be assigned into either the cohort of vaccinated or the cohort of unvaccinated health workers at the beginning of the follow-up period.

Vaccination data will be extracted from hospital records for the period of interest.

A database will be created with an identification code for each participant deriving from the tax code that will be unique but anonymous with the indication of the professional category. Sociodemographic data (i.e., age and sex) was retrieved from the employee tax code. Staff occupation information (i.e., physicians, nurses, and other health workers) will be obtained from the hospital human resources department.

The date of the first vaccination, the date of the second dose, batch numbers of the two doses, and the reason for the drop out of the second dose will be cataloged.

The data concerning positive swab results (i.e., validation date and type of swab) will be extracted through the hospital information systems. Information for adverse drug reactions will be retrieved from the national pharmacovigilance network for FPG Effectiveness of BNT162b2 vaccine against the transmission of SARS-CoV-2 will be measured. In particular, a vaccine breakthrough infection is defined as the detection of SARS-CoV-2 RNA or antigen, confirmed by a subsequent PCR test in a respiratory specimen collected from a person ≥14 days after they have completed all recommended doses of a European Medicines Agency-authorized COVID-19 vaccine The analysis of the vaccine safety among the health workers vaccinated during the vaccination campaign at FPG will be performed on the suspected adverse drug reactions spontaneously reported by the vaccination hub's team or HCWs retrieved from the national pharmacovigilance network (RNF). For the analysis, we consider the following: number of cases, demographic characteristic of the patients, seriousness, and symptoms reported. The terms for adverse reactions were coded as Preferred Terms (PT), according to the Medical Dictionary for Regulatory Activities (MedDRa), version 24.0.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers (aged ≥18 years) working at hospital sites who could provide written informed consent and who completed the immunization program with the administration of the second dose after approximately 21 days from the first dose at the FPG will be included

Exclusion Criteria:

* Participants were excluded from this analysis if they either will have a positive PCR test after 31 December 2020 and had clinical contraindications to the administration of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees of Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Sampling Method: Probability Sample
Enrollment: 6649 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Vaccine Effectiveness | 3 months
  BNT162b2 COVID-19 Vaccine effectiveness is interpreted as the proportionate reduction in disease attack rate among the vaccinated group
Vaccinese safety | 3 months
  Regarding the safety analysis of BNT162b2 COVID-19 Vaccine, the results of vaccine safety were descriptive in nature. Categorical data are presented as absolute and relative number of patients. For continuous data, mean and standard deviation (SD) or median with interquartile range (i.e., 1st quartile and 3rd quartile) was used, depending on its distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No